CLINICAL TRIAL: NCT03471585
Title: The Effects of Δ⁹-Tetrahydrocannabinol on the Retrieval of Emotional Memories
Brief Title: Effects of THC on Emotional Memory Retrieval
Acronym: TARE
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB16-1132
Record Dates: First submitted 2018-03-07; First posted 2018-03-20 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2018-03

CONDITIONS: Healthy
Keywords: THC; adult
MeSH Terms: interventions — Dronabinol; Glucose

STUDY DESIGN:
Intervention Model Description: Half of the participants will receive placebo during the second session in the first experimental arm and THC during the second session in the second experimental arm. The other half of participants will receive THC during the second session in the first experimental arm and placebo during the second session in the second experimental arm.
Who Masked: Participant, Investigator
Masking Description: A lab member that knew the design of the study but was not running participants sorted placebo and THC capsules into bags labeled "first capsule and "second capsule" for each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo oral capsule (Placebo Comparator): Participants came in for the first session that involved encoding emotional pictures and lists of semantically related words (Deese-Roediger-McDermott or DRM task; a false memory task). Forty-eight hours later, participants received a placebo capsule (dextrose) and waited 2 hours Participants were monitored for the next 2 hours including physiological and subjective measures every 30 minutes. After 2 hours, participants' memory for the emotional stimuli and DRM stimuli was tested. Participants then encoded object stimuli overlaid onto scenes followed by a working memory test with simple color squares. After the memory tests and 3.5 hours post-capsule, if participants' physiological and subjective measures had returned to baseline, they were allowed to leave. Forty-eight hours later, memory for the object-scene stimuli was tested. Other than the capsule, this arm was identical to the THC arm.
  Interventions: Drug: Placebo oral capsule
- THC (Experimental): Participants came in for the first session that involved encoding emotional pictures and lists of semantically related words (Deese-Roediger-McDermott or DRM task; a false memory task). Forty-eight hours later, participants received a placebo capsule (dextrose) and waited 2 hours Participants were monitored for the next 2 hours including physiological and subjective measures every 30 minutes. After 2 hours, participants' memory for the emotional stimuli and DRM stimuli was tested. Participants then encoded object stimuli overlaid onto scenes followed by a working memory test with simple color squares. After the memory tests and 3.5 hours post-capsule, if participants' physiological and subjective measures had returned to baseline, they were allowed to leave. Forty-eight hours later, memory for the object-scene stimuli was tested. Other than the capsule, this arm was identical to the placebo arm.
  Interventions: Drug: THC

INTERVENTIONS:
Drug: THC — A capsule that contains 15 mg of THC as well as dextrose filler administered 2 hours prior to memory testing.
  Other Names: Marinol
  Arms: THC
Drug: Placebo oral capsule — A capsule that contains only dextrose filler administered 2 hours prior to memory testing.
  Other Names: Dextrose
  Arms: Placebo oral capsule

SUMMARY:
The main purpose of this study was to examine the effects of THC on the retrieval of emotional and neutral memories in healthy young adults. Secondary experiments included the effects of THC on the encoding of object and scene stimuli and a novel working memory task.

DETAILED DESCRIPTION:
Here, the investigators aimed to investigate the effects of THC (15 mg) on the retrieval of negative, neutral, and positive memories. The study used a placebo-controlled, within-subjects, crossover design with 24 participants. In each experimental arm, participants attend a session to encode stimuli, a second session 48 hours later in which their memories are tested for the stimuli from the first session followed by the encoding of object-scene stimuli and a working memory test, and a third session 48 hours later in which memory for the object-scene stimuli is tested. In the second session, two hours prior to memory testing, THC or placebo is administered. On the first and second sessions subjects complete mood questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* 4-100 lifetime cannabis occasions

Exclusion Criteria:

* Current Axis I DSM-IV disorder, including substance dependence, current use of >5 cigarettes per day, history of psychosis or mania, less than a high school education, lack of English fluency, a body mass index outside 19-33 kg/m2, high blood pressure (>140/90), abnormal electrocardiogram, daily use of any medication other than birth control, pregnancy, or lactating.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2017-10-04 (Actual); Study Completion 2017-10-04 (Actual)

PRIMARY OUTCOMES:
Emotional Memory | Two hours after placebo/THC administration.
  Hit and false alarm rates for negative, neutral, and positive picture stimuli
DRM Memory | Two and a half hours after placebo/THC administration.
  Hit and false alarm rates for the DRM task
Object Memory | 48 hours after placebo/THC administration.
  Hit and false alarm rates for object stimuli on the same or different encoding scenes

SECONDARY OUTCOMES:
Addiction Research Centre Inventory Marijuana Scale | Assessed just prior to placebo/THC administration and then 30 minutes, 60 minutes, 90 minutes, and 115 minutes after placebo/THC administration.
  The Addiction Research Centre Inventory (ARCI; Martin, Sloan, Sapira, & Jasinski, 1971) measures drug-specific effects on a 56-item true-false questionnaire. For this study, the investigators report the composite score of 12 questions that make up the marijuana scale (Chait, Fischman, & Schuster, 1985).
Visual Analog Scales | Assessed just prior to placebo/THC administration and then 30 minutes, 60 minutes, 90 minutes, and 115 minutes after placebo/THC administration.
  The Visual Analog Scales (VAS; Folstein & Luria, 1973) is composed of thirteen adjectives used to assess individual dimensions of subjective mood - anxious, stimulated, sedated, elated, insightful, sociable, confident, lonely, playful, dizzy, loving, friendly, and restless, rated on a sliding scale from 'not at all' to 'extremely.'
Drug Effects Questionnaire | Assessed just prior to placebo/THC administration and then 30 minutes, 60 minutes, 90 minutes, and 115 minutes after placebo/THC administration.
  The Drug Effects Questionnaire (DEQ; Morean et al., 2013) is composed of five questions concerning current drug effects - how much participants feel a drug effect, like the effect, dislike the effect, feel high, and want more of the drug, rated on a sliding scale from 'not at all/neutral' to 'very much.'
Physiological Measure 1 | Assessed just prior to placebo/THC administration and then 30 minutes, 60 minutes, 90 minutes, and 115 minutes after placebo/THC administration.
  Heart rate
Physiological Measure 2 | Assessed just prior to placebo/THC administration and then 30 minutes, 60 minutes, 90 minutes, and 115 minutes after placebo/THC administration.
  Blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Harriet de Wit, PhD, Principal Investigator — University of Chicago; David A Gallo, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators have shared all of the data to https://osf.io/e6b5k/
Time Frame: The data is already available.
Access Criteria: Open to anyone.
URL: https://osf.io/e6b5k/

REFERENCES:
- [Derived] Doss MK, Weafer J, Gallo DA, de Wit H. Delta9-Tetrahydrocannabinol During Encoding Impairs Perceptual Details yet Spares Context Effects on Episodic Memory. Biol Psychiatry Cogn Neurosci Neuroimaging. 2020 Jan;5(1):110-118. doi: 10.1016/j.bpsc.2019.08.007. Epub 2019 Aug 30. PMID 31668830
- [Derived] Doss MK, Weafer J, Gallo DA, de Wit H. Delta9-Tetrahydrocannabinol at Retrieval Drives False Recollection of Neutral and Emotional Memories. Biol Psychiatry. 2018 Nov 15;84(10):743-750. doi: 10.1016/j.biopsych.2018.04.020. Epub 2018 May 9. PMID 29884456